CLINICAL TRIAL: NCT03042663
Title: Effect of Stellate Ganglion Block on Blood Flow in the Cannulated Radial Artery in Septic Shock Patients on Vasopressors, A Feasibility Study
Brief Title: Effect of Stellate Ganglion Block on Blood Flow in the Cannulated Radial Artery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eslam Ayman Mohamed Shawki (Other)
Responsible Party: Sponsor-Investigator, Eslam Ayman Mohamed Shawki, Lecturer of anesthesia, SICU & Pain Management, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: StArt
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Stellate Ganglion Block; Radial Artery Cannulation
Keywords: stellate ganglion block; arterial cannula; ischemia; septic shock
MeSH Terms: conditions — Ischemia; Shock, Septic

STUDY DESIGN:
Intervention Model Description: The study will recruit septic shock patients with hemodynamic instability on vasopressor support and on direct arterial blood pressure monitoring through a radial arterial cannula that is not older than 12 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): In patients meeting the inclusion criteria and with absence of any exclusion criteria, and after taking PI and Doppler Blood flow values hourly for 3 hours (control values), the procedure for administering the USG Stellate ganglion block on the side of the arterial cannula will be started
  Interventions: Procedure: USG stellate ganglion block

INTERVENTIONS:
Procedure: USG stellate ganglion block — After verification of proper needle position and aspiration to exclude vascular spread, 1mL of the injectate will be injected to see proper tissue spread as well as patient response. After one minute the remaining volume will be injected under real time ultrasound imaging.

SUMMARY:
To evaluate the value of US-guided Stellate ganglion block for improving radial arterial blood flow and peripheral perfusion in Septic shock patients on vasopressor support with an indwelling radial arterial cannula, which can result in reduced incidence premature failure of the catheter (due to vasospasm or thrombosis) and incidence of ischemic complications in the cannulated arm.

DETAILED DESCRIPTION:
Radial artery cannulation is a well-established procedure in the ICU, especially in critically ill hemodynamically unstable patients. The first description of arterial cannulation in humans dates back to 1856, when the blood pressure was measured int the femoral artery. It can be used for continuous blood pressure monitoring, obtaining func¬tional hemodynamic parameters derived from the arterial waveform, to predict the physiologic response to fluid resuscitation and also for blood sampling.

The most common complications for the procedure are temporary radial artery occlusion (19.7%), in addition to hematoma (14.4%), infection at the arterial site (0.72%), hemorrhage (0.53%) or bacteremia (0.13%), pseudoaneurysm (0.09%) and finally ischemic damage (0.09%). Larger catheter diameter, presence of vasospasm, female sex (probably related to smaller vessel diameter) increase the risk of ischemic complications. Inadequate experience (high number of attempts, multiple arterial sticks and hematoma formation) can also increase the complication rate.

In a recent study by Numaguchi et al, they found that radial artery cannulation decreases the distal arterial blood flow measured by power Doppler ultrasound. In another study by Kim et al, they found that after radial artery cannulation ulnar artery diameters were significantly increased (compensatory) and radial artery diameters were decreased after cannulation compared with pre-cannulation values, then returned to pre-cannulation values 5 min after cannulation. They detected radial artery vasospasm in 12 patients with 20-G cannulas used (31.5%) and in 2 patients with 22-G cannulas used (5.3%) (p < 0.05), which was observed immediately after cannulation, and had mostly disappeared after 5 min. There was no data regarding the follow up of the patients afterwards. In both studies the subjects were not critically ill patients (and not on vasopressors).

Peripheral limb ischemia in ICU patients can be the result of iatrogenic injury, thrombotic complications or hypoperfusion related to the underlying disease state. The patients at greatest risk for acute ischemia are those with underlying peripheral artery disease (PAD), but limb ischemia can also be the consequence of embolism, injury, dissection, or severe vasoconstriction, even in the absence of preexisting occlusive disease. Repeated arterial punctures may result in extensive hematoma formation and arterial spasm, The thick muscular coat and abundance of alpha adrenoreceptors make it prone to develop spasm when traumatized. Attempts to control bleeding following cannulation through local hemostasis only complicate matters. While, normally, the likelihood of serious ischemia is minimized by the presence of the palmar arterial arch.

The use of vasopressors especially nor-epinephrine with its potent α1-adrenergic receptor agonist activity can aggravate the condition more. We didn't find in the literature any reliable data regarding the effect of using vasopressors (particularly nor-epinephrine) in any dosage on the incidence of peripheral arterial vasospasm or ischemic complications following arterial cannulation. But there were mixed case reports linking both or one of them: high dose vasopressors and arterial cannulation, to ischemic complications. Such as developing peripheral gangrene after starting high dose vasopressors, or developing complex regional pain syndrome (CRPS) following radial artery cannulation.

It is believed that blocking the Stellate ganglion with Local anesthetics can interfere with the sympathetic out flow to the upper limb resulting in abolishing its vasoconstrictor action on the arteries thus decreasing arterial spasm and promoting better blood flow in the peripheral circulation.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-80 years.
* Septic shock patients on vasopressor support (Nor-epinephrine or epinephrine).
* Presence of an indication for an arterial cannula.

Exclusion Criteria:

* Coagulopathies (with prothrombin concentration less than 60% or international normalized ratio INR more than 1.5)
* In-ability to postpone anti-coagulation medications.
* Infection or injury or a lesion at the block site.
* Suspected cervical vertebral column injury necessitating using a neck collar.
* Bradycardia with heart rate less than 60 beat per minute.
* A compromised lung on the contralateral side of the arterial cannula (Pneumothorax, hemothorax or Pneumonectomy).
* Recent cardiac insult (cardiogenic shock) (Due to blockage of the sympathetic cardiac accelerator fibers by the block).
* Traumatic vascular injuries or operative interventions (Surgical harvesting) involving arteries of the upper limb on either side.
* Peripheral vascular disease, atherosclerosis, atrial fibrillation, previous history of ischemic injuries, hypercoagulable syndromes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-10-04 (Estimated)

PRIMARY OUTCOMES:
change in Perfusion Index (PI) | After 30 minutes then every hour for 6 hours
  change in Perfusion Index (PI) in the cannulated limb before and after the Stellate ganglion block.

SECONDARY OUTCOMES:
Perfusion Index (PI) after cannulation | 3 hours
  Perfusion Index (PI) values bilaterally after radial arterial cannulation
Perfusion Index (PI) after Stellate ganglion block | 6 hours
  Perfusion Index (PI) values bilaterally after Stellate ganglion block in the cannulated side.
Doppler Blood flow values after cannulation | 3 hours
  Doppler Blood flow values in the both Radial arteries after cannulation of one of them.
Doppler Blood flow after Stellate ganglion block | 6 hours
  Doppler Blood flow values in the both Radial arteries after Stellate ganglion block in the cannulated side.
Vasopressor drug dose | 6 hours
  Doses of vasopressor drugs used.
Incidence of complications | 6 hours
  Incidence of complications related to the Stellate ganglion block (Hematoma, Intravascular injection, Intrathecal injection, pneumothorax).
Incidence of ischemic complications | 6 hours
  Incidence of ischemic complications related to the arterial cannula (Unilateral) or Vasopressors and general condition of the patient (Bilateral) (changes in the form of either color changes or definite gangrene).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo University teaching hospitals (Kasr Alainy), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Gershengorn HB, Garland A, Kramer A, Scales DC, Rubenfeld G, Wunsch H. Variation of arterial and central venous catheter use in United States intensive care units. Anesthesiology. 2014 Mar;120(3):650-64. doi: 10.1097/ALN.0000000000000008. PMID 24424071
- [Background] Scheer B, Perel A, Pfeiffer UJ. Clinical review: complications and risk factors of peripheral arterial catheters used for haemodynamic monitoring in anaesthesia and intensive care medicine. Crit Care. 2002 Jun;6(3):199-204. doi: 10.1186/cc1489. Epub 2002 Apr 18. PMID 12133178
- [Background] Glockner E, Harych H. [Guidelines for planning concerning physicians and stomatologists up to 1980]. Z Gesamte Hyg. 1970 Oct;16(10):811-22. No abstract available. German. PMID 5516161
- [Background] Kim SY, Lee JS, Kim WO, Sun JM, Kwon MK, Kil HK. Evaluation of radial and ulnar blood flow after radial artery cannulation with 20- and 22-gauge cannulae using duplex Doppler ultrasound. Anaesthesia. 2012 Oct;67(10):1138-45. doi: 10.1111/j.1365-2044.2012.07235.x. Epub 2012 Jul 16. PMID 22804619
- [Background] Lazaro RP. Complex regional pain syndrome and acute carpal tunnel syndrome following radial artery cannulation: a neurological perspective and review of the literature. Medicine (Baltimore). 2015 Jan;94(3):e422. doi: 10.1097/MD.0000000000000422. PMID 25621693
- [Background] Rasmy I, Mohamed H, Nabil N, Abdalah S, Hasanin A, Eladawy A, Ahmed M, Mukhtar A. Evaluation of Perfusion Index as a Predictor of Vasopressor Requirement in Patients with Severe Sepsis. Shock. 2015 Dec;44(6):554-9. doi: 10.1097/SHK.0000000000000481. PMID 26529657
- [Background] Yamazaki H, Nishiyama J, Suzuki T. Use of perfusion index from pulse oximetry to determine efficacy of stellate ganglion block. Local Reg Anesth. 2012;5:9-14. doi: 10.2147/LRA.S30257. Epub 2012 Mar 13. PMID 22915896